CLINICAL TRIAL: NCT03121703
Title: Main Researcher for Effects of Lumbar Stabilization Exercise on Transversus Abdominis Muscle Activation Capacity and Function in Chronic Low Back Pain Patients
Brief Title: The Effects of Lumbar Stabilization Exercise on Transversus Abdominis Muscle Activation Capacity and Function in Chronic Low Back Pain Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Do hyun Kim, Principal Investigator, Inje University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: InjeU 1
Record Dates: First submitted 2017-04-12; First posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lumbar stabilization exercises group (Experimental): diverse lumbar stabilization exercises
  Interventions: Other: lumbar stabilization exercise
- trunk muscle strengthening exercise (Other): trunk muscle strengthening exercise
  Interventions: Other: trunk muscle strengthening exercise

INTERVENTIONS:
Other: lumbar stabilization exercise — lumbar stabilization exercise
  Arms: lumbar stabilization exercises group
Other: trunk muscle strengthening exercise — trunk muscle strengthening exercise
  Arms: trunk muscle strengthening exercise

SUMMARY:
Purpose: The purpose of this study is to investigate the effects of lumbar stabilization exercises on pain intensity, transversus abdominis muscle (TrA) activation capacity, functional disability, and TrA thickness in patients with chronic low back pain (CLBP). Subjects: The subjects of this study were 30 CLBP patients. Methods: The experimental group performed diverse lumbar stabilization exercises in different postures, and the control group conducted an ordinary trunk muscle strengthening exercise. Results: There were significant differences in pain intensity, TrA activation capacity, functional disability, and TrA thickness between before and after the intervention in both groups. Significant differences between the two groups were shown in the pain intensity, TrA activation capacity, and functional disability after the intervention. However, there were no significant differences between the two groups in TrA thickness. Conclusion: Lumbar stabilization exercises in different postures could reduce pain, functional disability, and increase TrA activation capacity and thickness in CLBP patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who felt low back pain

Exclusion Criteria:

* Orthopedic surgery within 6 months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2017-05-30 (Estimated); Study Completion 2017-06-30 (Estimated)

PRIMARY OUTCOMES:
transverse abdominis thickness | 1 year
  ultrasound image for measuring transverse abdominis thickness